CLINICAL TRIAL: NCT01583803
Title: Investigation of the Sex Differences in Oral Microbiota and Their Effect on Circulating Nitrite Levels
Brief Title: Sex Differences in Oral Bacteria
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Queen Mary University of London (Other)
Collaborators: King's College London (Other)
Responsible Party: Principal Investigator, Amrita Ahluwalia, Professor of Vascular Pharmacology, Queen Mary University of London
Other Study IDs: 12/LO/0108
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, saliva and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Males
- Females

SUMMARY:
Females have a lower incidence of hypertensive and cardiovascular disorders that may relate to differences in nitrogen oxides in the blood and saliva. Some nitrogen oxides are recycled with the help of oral bacteria to nitric oxide which is protective against vascular disorders. This study will test the hypothesis that females have different numbers and species of these nitrogen-oxide reducing bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18-45 who have volunteered themselves and are willing to sign the consent form

Exclusion Criteria:

1. Healthy subjects unwilling to consent
2. History of hypertension, diabetes or hypertensive on BP measurement
3. Pregnant, or any possibility that a subject may be pregnant unless in the latter case a pregnancy test is performed with a negative result
4. History of any serious illnesses, including recent infections or trauma
5. Subjects taking systemic medication (other than the oral contraceptive pill)
6. Subjects with self-reported use of mouthwash or tongue scrapes
7. Subjects with recent or current antibiotic use (within 3 months)
8. Subjects with a history, or recent treatment of (within last 3 months) of any oral condition (excluding caries), including gingivitis, periodontitis and halitosis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-01 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Bacterial species identification | At baseline

SECONDARY OUTCOMES:
Bacterial count | At baseline
Blood pressure | At baseline
Nitrogen oxide levels in biological fluids | At baseline
Oral nitrate reduction | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Ahluwalia, PhD, Principal Investigator — Queen Mary University London
Locations (1):
- William Harvey Heart Centre, London, United Kingdom

REFERENCES:
- [Background] Kapil V, Milsom AB, Okorie M, Maleki-Toyserkani S, Akram F, Rehman F, Arghandawi S, Pearl V, Benjamin N, Loukogeorgakis S, Macallister R, Hobbs AJ, Webb AJ, Ahluwalia A. Inorganic nitrate supplementation lowers blood pressure in humans: role for nitrite-derived NO. Hypertension. 2010 Aug;56(2):274-81. doi: 10.1161/HYPERTENSIONAHA.110.153536. Epub 2010 Jun 28. PMID 20585108
- [Derived] Kapil V, Rathod KS, Khambata RS, Bahra M, Velmurugan S, Purba A, S Watson D, Barnes MR, Wade WG, Ahluwalia A. Sex differences in the nitrate-nitrite-NO* pathway: Role of oral nitrate-reducing bacteria. Free Radic Biol Med. 2018 Oct;126:113-121. doi: 10.1016/j.freeradbiomed.2018.07.010. Epub 2018 Jul 20. PMID 30031863